CLINICAL TRIAL: NCT01543165
Title: A Single Center, Prospective Randomized Double-blind Trial: Efficacy of Nefopam and Morphine in Balanced Analgesia for Acute Ureteric Colic
Brief Title: Efficacy of Nefopam and Morphine in Balanced Analgesia for Acute Ureteric Colic
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Pharmbio Korea (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B-1112/141-011
Record Dates: First submitted 2012-02-27; First posted 2012-03-02 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Renal Colic
Keywords: Renal colic; Analgesia; Nefopam; Ketorolac
MeSH Terms: conditions — Renal Colic; Agnosia | interventions — Ketorolac; Morphine; Analgesia; Analgesics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Group 1 (Experimental): Sequential intravenous administration of ketorolac and nefopam
  Interventions: Drug: Ketorolac and nefopam balanced analgesia
- Group 2 (Active Comparator): Sequential intravenous administration of ketorolac and morphine
  Interventions: Drug: Balanced analgesia using ketorolac and morphine
- Group 3 (Placebo Comparator): Intravenous administration of ketorolac
  Interventions: Drug: Pain control with single analgesics (ketorolac)

INTERVENTIONS:
Drug: Ketorolac and nefopam balanced analgesia — Sequential intravenous administration of ketorolac and nefopam
  Arms: Group 1
Drug: Balanced analgesia using ketorolac and morphine — Sequential intravenous administration of ketorolac and morphine
  Arms: Group 2
Drug: Pain control with single analgesics (ketorolac) — This arm do not use balanced analgesia. Instead, ketorolac IV administration followed by 50cc normal saline administration (for blinding) will be used in this group.
  Arms: Group 3

SUMMARY:
This study is to see whether the combination regimen of ketorolac and nefopam is superior to that of ketorolac and morphine in controlling ureter stone-related acute flank pain.

DETAILED DESCRIPTION:
The balanced analgesia regimen using both ketorolac and morphine is the most effective choice in controlling urolithiasis related acute pain. Previous animal and human studies reported that combination regimen of ketoprofen and nefopam showed synergistic effect in pain control. We hypothesized that using nefopam instead of morphine for ketorolac based combination analgesia will produce similar pain reduction without causing opioid-related side effect.

ELIGIBILITY:
Inclusion Criteria:

* Acute flank with visual analog pain scale score equal or more than 5
* and most possible diagnosis after initial clinical exam is acute renal colic

Exclusion Criteria:

* Pregnant or lactating women
* Patients whose use of any of the study drugs is contraindicated
* Patients with documented renal or hepatic failure or those with clinical findings suggesting the diagnoses
* Recent episode of acute myocardial infarction or patients with significant heart failure
* Patients with documented gastric/duodenal ulcer or those with clinical findings suggesting the diagnoses
* Patients with bleeding tendency
* Patients who have history of any seizure
* Patients with documented organic brain injury
* Patients taking warfarin
* Patients whose primary diagnosis is not renal colic

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 111 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Amount of pain reduction by visual analog pain scale | At 30 and 60 minutes after primary study drug administration

SECONDARY OUTCOMES:
Additional analgesia requested by enrolled patients | At 30 and 60 minutes after primary study drug administration

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Kyeongi-do, South Korea